CLINICAL TRIAL: NCT02178449
Title: The Effect of Dexamethasone Used Together With Low Volume Ropivacaine in a Single Shot Interscalene Block on the Pain Free Time Experienced by the Patient
Brief Title: Prolongation of Pain Free Time by the Use of Dexamethasone in Peripheral Nerve Blockade
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Landesklinikum Sankt Polten (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DEXATrial1; GS4-EK-2/304-2013 (Other: Ethics commission of lower austria)
Record Dates: First submitted 2014-05-26; First posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Interscalene Block; Shoulder Arthroscopy; Dexamethasone; Low Volume Regional Anesthesia
MeSH Terms: interventions — dexamethasone acetate; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum (Experimental): Dexamethasone and Ropivacaine
  Interventions: Drug: Dexamethasone acetate; Drug: Ropivacaine
- Placebo (Active Comparator): Ropivacaine and Saline
  Interventions: Drug: Placebo; Drug: Ropivacaine

INTERVENTIONS:
Drug: Dexamethasone acetate
  Arms: Verum
Drug: Placebo
  Arms: Placebo
Drug: Ropivacaine

SUMMARY:
The main aim of the study is to investigate the proven effect of dexamethsone on the duration of the interscalene block. The investigators try to define optimal dose and volume for ropivacaine, when used together with dexamethsone. The current literature uses often very high volumes of ropivacain when used together with dexamethasone. The investigators try to research the effect of using dexamethsone together with low volume, high concentration ropivacaine for interscalene blockade. The investigators' hypothesis is that dexamethasone has an positive effect on the pain free after used together with ropivacaine at the scalene block.

ELIGIBILITY:
Inclusion Criteria:

* atroscopy of the shoulder
* repair of the RM

Exclusion Criteria:

* patient under 18 years
* patient is fertile
* chronic opiat use more than 30mg oxycodone per day
* operations at the shoulder that involves the bone
* usage of cortisone for more than 2 weeks
* risk greater as asa III
* damage to nerves
* neuropathy at the target arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-04 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Pain free time measured by the duration between block and the point at which the patient is asking for painkillers | Patients will be followed during their stay at the hospital, which will be normally around 24 to 48 hours.

SECONDARY OUTCOMES:
Visual Rating Scale for Pain at Movement and Rest | Measured 10 hours after the intervention

OTHER OUTCOMES:
Patient satisfaction | 1 day, when the patient leaves the hospital
  Measured by a validated questionary

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hörmann, MD, Study Director — Landesklinikum Sankt Polten
Locations (1):
- Landesklinikum Sankt Pölten, Sankt Pölten, Lower Austria, Austria